CLINICAL TRIAL: NCT02018874
Title: A Phase Ib, Open-label, Dose Escalation Study of the Safety, Tolerability and Efficacy of LY2780301 (a p70/AKT Inhibitor) in Combination With Gemcitabine in Patients With Advanced or Metastatic Cancer
Brief Title: A Phase Ib Study of the Safety, Tolerability and Efficacy of LY2780301 in Combination With Gemcitabine
Acronym: INPAKT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-000671-33; 2013/1975 (Other: CSET number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-23 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Solid Tumors and Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2780301 (Experimental)
  Interventions: Drug: LY2780301; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2780301 — LY2780301 will be given orally Q.D. at different dose levels. Because of a favourable safety profile, the different dose levels will be as follow :
  * Dose level -1: 300 mg Q.D.
  * Dose level -0.5: 400 mg Q.D.
  * Dose level 1: 400 mg Q.D.
  * Dose level 1.5: 500 mg Q.D.
  * Dose level 2 : 500 mg Q.D.
Drug: Gemcitabine — The dose level of Gemcitabine will be fixed (1000 mg/m2). Gemcitabine will be administered over a 30 minutes infusion.

SUMMARY:
In the First-in-Human, JWAA trial, the LY2780301 displayed a favourable safety profile, a high pharmacokinetic exposure and the ability to decrease pS6. LY2780301 has shown synergistic activity in combination with targeted agents or chemotherapy including gemcitabine. We propose herein to combine LY2780301 with gemcitabine and to treat different tumor types with molecular alterations. This may validate the anti-tumor activity of the LY2780301 and it will increase our knowledge regarding molecular predictors of its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Dose Escalation portion (Part 1): have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic disease (including Non-Hodgkin's Lymphoma) with selected molecular alterations and for which no proven effective therapy exists. ;
2. Dose Confirmation portion (Part 2): have histological or cytological evidence of cancer (solid tumor or Non-Hodgkin's Lymphoma) that is advanced and/or metastatic disease:

   * Cohort A: Up to 20 patients of any histological type (solid tumor or Non-Hodgkin's Lymphoma) with selected molecular alterations
   * Cohort B: Up to 12 patients with ovarian cancer and with selected molecular alterations 1.1 (Appendix 4) for solid tumors or by the Revised Response Criteria for Malignant Lymphoma

Dose Confirmation portion:

* Measurable disease as defined by RECIST 1.1 for solid tumors (Appendix 4) except ovarian cancer or
* Response Criteria for Patients with Ovarian Cancer Who Have Evaluable but Non-Measurable Disease (Appendix 5) or
* Revised Response Criteria for Non-Hodgkins Lymphoma (Appendix 6) [4] Are >/=18 years of age ; [5] Written informed consent ; [6] Have adequate organ function including:

  * Hematologic: absolute neutrophil count (ANC) >/=1.5 x 109/L, platelets

    >/=100 x 109/L, and hemoglobin >/=9 g/dL.
  * Hepatic: bilirubin </=1.5 times upper limits of normal (ULN); alanine transaminase (ALT) and AST </=2.5 x ULN. (</=5 x ULN if the liver has tumor involvement).
  * Renal: Serum creatinine </=1.5 x ULN or calculated creatinine clearance >45 ml/min (MDRD) [7] ECOG performance status </= 1 ; [8] Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 2 weeks (3 weeks for myelosuppressive agents) prior to study enrolment and all prior treatment related toxicities must be CTCAE (Version 4.0) </= Grade 1 (except alopecia) at the time of enrolment. Patients with prostate cancers progressing under LHRH agonist therapy, may have that treatment continued while receiving study drug ; [9] Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 6 months following the last dose of study drug ; [10] Females with childbearing potential must have had a negative serum pregnancy test </= 14 days prior to the first dose of study drug ; [11] Have an estimated life expectancy >/=12 weeks ; [12] Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels ;

Exclusion Criteria:

[13] Any serious and/or unstable pre-existing medical conditions, psychiatric disorder, or other conditions that could, in the opinion of the investigator, interfere with subject's safety, obtaining informed consent or compliance to the study procedures ; [14] Have symptomatic CNS malignancy or symptomatic brain metastasis. Patients with treated CNS metastases are eligible provided their disease is radiographically stable and asymptomatic and they are not currently receiving corticosteroids. Screening of asymptomatic patients without history of CNS metastasis is not required ; [15] Have pre-existing not controlled cardiovascular disease (including acute coronary syndromes, unstable angina, coronary angioplasty, or stenting within the past 6 months) or any QTc prolongation (defined as a QTc interval > 480 ms according to Friedericia's correction) or other significant ECG abnormalities including 2nd degree AV block type II, 3rd degree AV block, or bradycardia (HR < 50 bpm), or any history of 2nd or 3rd degree block ; [16] Concomitant treatment prohibited in section 7.8 ; [17] Pregnancy and Breast Feeding ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 4 weeks
  Patients fulfilling the inclusion criteria will be enrolled in successive cohorts of 3 to 6 patients. If no DLT is observed during the first 4 weeks of study treatment in 3 patients, the dose of LY2780301 will be escalated to the dose level (DL) immediately above. If One DLT is observed among 3 patients, the cohort will be expanded to 6 evaluable patients. If two patients out of 3 or 2 /6 patients experience a DLT, the dose will be considered intolerable and the DL immediately below will be further explored. The recommended phase II dose (RP2D) will be the highest DL in which no more than 1/6 patients experiences a DLT. If no DLT is observed at the highest planned DL, this DL will be deemed the RP2D. Intermediate DLs could be added, if clinically relevant.
Efficacy | Assessed every 8 weeks from inclusion until progression up to 5 months
  * Solid Tumors: Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
  * Non-Measurable Ovarian Cancer: Response Criteria for Patients with Ovarian Cancer Who Have Evaluable but Non-Measurable Disease
  * Non-Hodgkin Lymphoma: the Revised Response Criteria for Malignant Lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Jean Charles Soria, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Angevin E, Cassier PA, Italiano A, Goncalves A, Gazzah A, Terret C, Toulmonde M, Gravis G, Varga A, Parlavecchio C, Paci A, Poinsignon V, Soria JC, Drubay D, Hollebecque A. Safety, tolerability and antitumour activity of LY2780301 (p70S6K/AKT inhibitor) in combination with gemcitabine in molecularly selected patients with advanced or metastatic cancer: a phase IB dose escalation study. Eur J Cancer. 2017 Sep;83:194-202. doi: 10.1016/j.ejca.2017.06.036. Epub 2017 Jul 24. PMID 28750271
- See also: Related Info — http://www.gustaveroussy.fr/fr/essai